CLINICAL TRIAL: NCT02770365
Title: Comparative Safety and Efficacy of Two Treatments in the Treatment of Vulvar and Vaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Collaborators: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-15-007
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Atrophy
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product (Experimental): estradiol cream
  Interventions: Drug: estrace cream (Perrigo)
- Reference Product (Active Comparator): estradiol cream
  Interventions: Drug: estrace cream (Reference)
- Placebo product (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: estrace cream (Perrigo)
  Other Names: Perrigo product
  Arms: Test Product
Drug: estrace cream (Reference)
  Other Names: Reference Listed Drug product
  Arms: Reference Product
Drug: Placebo cream
  Arms: Placebo product

SUMMARY:
To compare safety and efficacy of Perrigo's drug product compared to an FDA approved drug product in the treatment of vulvar and vaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal female and otherwise healthy, 30 - 75 years of age.
* ≤ 5% superficial cells on vaginal smear cytology at Visit 1/Screening.
* vaginal pH > 5.0 at Visit 1/Screening
* Have at least one self-assessed moderate to severe symptom of Vulvar and Vaginal Atrophy identified by the subject as being the most bothersome
* For women with an intact uterus, vaginal ultrasonography confirmation at Visit 1/Screening of an inactive endometrial lining with an endometrial thickness less than 4 mm.
* Systolic blood pressure no greater than 150 mm Hg and diastolic blood pressure no greater than 90 mm Hg at Visit 1/Screening and at Visit 2/Randomization

Exclusion Criteria:

* Undiagnosed vaginal bleeding or a history of significant risk factors for endometrial cancer.
* Known, suspected, or history of cancer of the breast or mammogram indicating any abnormalities or subject has a history of cervical cancer.
* Vaginal ultrasonography for all women with an intact uterus confirming endometrial thickness of 4mm or more
* History of hypersensitivity or allergy to estradiol or any of the other study medication ingredients.
* Known or suspected estrogen-dependent neoplasia.
* Has deep vein thrombosis, pulmonary embolism or history of these conditions.

  • Subject has active arterial thromboembolic disease (e. g. stroke, myocardial infarction) or history of these conditions.
* Known acute or chronic hepatic disease or dysfunction

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Clinical Trials, LLC, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: estradiol cream
  estrace cream (Perrigo)
- Reference Product: estradiol cream
  estrace cream (Reference)
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo Product
Started | 277 | 279 | 139
Completed | 272 | 275 | 139
Not Completed | 5 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo Product | Total
Number analyzed (Participants) | 275 | 277 | 139 | 691
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (6.35) | 59.9 (6.31) | 59.2 (6.06) | 59.9 (6.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 277 | 139 | 691
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 59 | 29 | 143
  Not Hispanic or Latino | 220 | 218 | 110 | 548
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 5 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 33 | 35 | 25 | 93
  White | 233 | 235 | 114 | 582
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Identified as Responders
Description: A responder is a subject meeting specific vaginal cytology criteria AND a vaginal pH < 5.0 with a change from Visit 1 of at least 0.5.
Time Frame: Day 8
Population: Per protocol population
Measure: Number; unit: percentage of responders
Arm/Group | Test Product | Reference Product | Placebo Product
Number analyzed (Participants) | 228 | 231 | 121
percentage of responders | 36.8 | 32.0 | 0.8
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — provides 85% power of success; Wald's method; Equivalence ratio = 1.14, 90% CI 2-sided [-2.92 to 12.53]

2. Secondary Outcome: Most Bothersome Symptom
Description: Percentage of subjects based on the improvement (change from Visit 2) of the Most Bothersome Symptom at Visit 3.
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 217 | 214
Participants | 116 | 123
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — the proportion of subjects with treatment success based on the improvement of the Most Bothersome Symptom (MBS) of vulvo-vaginal atrophy at Day 8; p = 0.05, Wald's method; equivalence ratio = 0.94, 90% CI 2-sided [-12.35 to 4.31]

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | Test Product | Reference Product | Placebo Product
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/279 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/277 | 0/279 | 0/139
Other Adverse Events (participants affected / at risk) | 0/277 | 0/279 | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's cannot disclose trial results under any circumstances.

DOCUMENTS (2):
  • Study Protocol (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT02770365/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT02770365/SAP_001.pdf